CLINICAL TRIAL: NCT06654154
Title: Vitamin B12: a Biological Marker of Systemic Disease or Infection Flare-up in Patients Treated with Tocilizumab?
Acronym: TOCI2C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RNI 2023 CLEMENT; 2023-A01673-42 (Other: ANSM)
Record Dates: First submitted 2024-03-20; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Level of Serum Vitamin B12 Level (in Pmol/L) If Relapse of (AI/ID) Under Tocilizumab; Level of Serum Vitamin B12 Level (in Pmol/L) If Infection Under Tocilizumab
Keywords: vitamin B12; Tocilizumabe; autoimmune desease; auto-inflammatory disease

STUDY DESIGN:
Intervention Model Description: Determination of serum level of vitamin B12 and data collection in a patient:
  * At study inclusion
  * If an infection or a AI/ID relapse is suspected
  * At remission in case if inclusion during AI/ID relapse
  * At tocilizumab initiation if happening along with inclusion
  * At Day 3 (+/-1) if an infection or AI/ID relapse is suspected and if the patient is hospitalized and if a blood test is realised
Masking Description: Each patient is his own witness to express the variation in the serum level of vitamin B12: this way we overcome individual variability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- study the variation in serum vitamin B12 level (Other): Each patient is his own witness to express the variation in the serum level of vitamin B12
  Interventions: Diagnostic Test: variation of serum level vitamine B12

INTERVENTIONS:
Diagnostic Test: variation of serum level vitamine B12 — There will be no specific visit to the study. Follow-up in consultation will be done by your referring doctor. A determination of the serum level of vitamin B12 will be carried out at inclusion, during a consultation where the pathology is in remission (during the classic assessment of follow-up under tocilizumab, left to the discretion of the patient's referring doctor. ). It will also be necessary to carry out, in addition to the classic assessment left to the discretion of the patient's doctor, a determination of the serum level of vitamin B12 in the event of clinical suspicion of infection or an outbreak of MAI/I.
  The determination of serum vitamin B12 requires the collection of an additional tube of 300 μl of venous blood but no additional venipuncture

SUMMARY:
Tocilizumab is a monoclonal antibody that acts as an IL-6 receptor antagonist It is responsible for a reduction in the hepatic synthesis of inflammatory proteins, including CRP (C-reactive protein).

Thus, the diagnosis of a relapse of the autoimmune or auto inflammatory disease (AI/ID) or an infection is made difficult in patients treated with tocilizumab and there is to date no marker of inflammation validated in patients receiving tocilizumab.

Vitamin B12 is an essential element that participates to haematopoiesis, myelin integrity, neuronal function and DNA synthesis. Vitamin B12 is carried by haptocorrin and transcobalamin II (TCII). Vitamin B12 increases in many pathological situations, including infections and AI/ID due to the increase of its transport proteins elevation (mostly transcobalamin II).

The sponsor did not find any study in the literature studying the level of vitamin B12 or TCII in patients taking tocilizumab. The sponsor also did not find any physiopathological argument in favor of an inhibition of TCII synthesis by tocilizumab.

As such, TCII dosage could be of interest, but the dosage is not available in routine whereas vitamin B12 dosage is available in every laboratory and is four times cheaper.

DETAILED DESCRIPTION:
The main objective is to study the variation in serum vitamin B12 level in case of clinical suspicion of AID/I flare or infection in patients treated with tocilizumab compared to the B12 level of the patient in remission period. , and excluding infection, under tocilizumab

Also, serum vitamin B12 will be measured during a biological assessment carried out either in the event of a suspected outbreak of MAI/I or infection, or in the event of remission (during the follow-up assessment carried out systematically in a patient on tocilizumab).

This determination of serum vitamin B12 will be carried out during a blood test carried out at the request of the patient's doctor.

The study will involve taking an additional tube of venous blood but will not result in additional venipuncture.

There will be no specific visit related to the study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patient with:

  * A diagnosis of rheumatoid arthritis according to ACR EULAR 2010 classification criteria
  * Or a diagnosis of polymyalgia rheumatica according to ACR EULAR 2012 classification criteria
  * Or a diagnosis of giant cell arteritis (with or without polymyalgia rheumatica associated) according to 2022 revised classification criteria
  * Or a diagnosis of systemic sclerosis according to ACR EULAR 2013 classification criteria
  * Or a diagnosis of Takayasu vasculitis according to ACR 2022 classification criteria
  * Or a diagnosis of Still disease according to Yamaguchi or Fautrel classification criteria
  * Or a diagnosis of VEXAS with UBA1 somatic mutation
  * Or a diagnosis of unclassified autoimmune or auto-inflammatory disease treated by tocilizumab
* Receiving intravenous or subcutaneous tocilizumab (treatment can be introduce before inclusion or started at the inclusion)
* Capable of giving informed consent
* Covered by a social protection system

Exclusion Criteria:

* Patient treated by oral or subcutaneous vitamin B12
* Pregnant or breastfeeding women
* Patient under guardianship or curatorship, deprived or liberty, placed under judicial protection
* Rejection to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Variationof serum level of vitamin B12 (pmol/L) between a clinical suspicion of relapse autoimmune or autoinflammatory desease (AI/ID) or infection and a remission state, in patients treated by tocilizumab. | - At study inclusion - During the 3 years of the patient's participation and if included during a remission, new sample in case of suspicion of new infection or recurrence of autoimmune or inflammatory disease - During the 3 years of the patient's par
  Percentage change of vitamin B12 serum level (pmol/L) between a remission state without infection ongoing and an relapse AI/ID or an infection.

SECONDARY OUTCOMES:
Description of distribution of patients according to occurrence infection or AI/ID desease. | from enrollment to the 3 years of the patient's participation
  Occurrence of infection or autoimmune-autoinflammory desease.
variation of serum vitamin B12 level (pmol/L) according the events | from enrollment to the 3 years of the patient's participation
  Percentage change of vitamin B12 serum level (pmol/L) between level in remission and level in relapse AI/ID or infection Percentage change of vitamin B12 serum level (pmol/L) between level at the start (J0) of relapse AI/ID or infection and at J3 of the start of relapse AI/ID or infection
variation of serum vitamin B12 level (pmol/L) according event under treatment | from enrollment to the 3 years of the patient's participation
  Percentage change of vitamin B12 serum level (pmol/L) under Tocilizumab between level in remission and level in relapse AI/ID or infection
variation of serum vitamin B12 level (pmol/L) according the duration of treatment by tocilizumab | from enrollment to the 3 years of the patient's participation
  Percentage change of vitamin B12 serum level (pmol/L) according the duration of treatment and occurrence of relapse of AI/ID or infection
  l
variation of serum vitamin B12 level (pmol/L) according Previous AI/ID treatment | from enrollment to the 3 years of the patient's participation
  According the previous treatment, percentage change of vitamin B12 serum level (pmol/L) at the inclusion
variation of serum vitamin B12 level (pmol/L) according patients characteristics | from enrollment to the 3 years of the patient's participation
  Percentage change of vitamin B12 serum level (pmol/L) according to sexe (women-man) Percentage change of vitamin B12 serum level (pmol/L) according to weight (kg) Percentage change of vitamin B12 serum level (pmol/L) according to age (years)
Comparaison of the level serum vitamin B12 level (pmol/L) in relapse AI/ID or infection with other inflammatory markers: | from enrollment to the 3 years of the patient's participation
  comparaison between the level vitamin B12 serum and the level of CRP (mg/L) and fibrogène (g/L) performed at the same time during study
variation of serum vitamin B12 level (pmol/L) according the way of tocilizumab administration | from enrollment to the 3 years of the patient's participation
  Percentage change of vitamin B12 serum level (pmol/L) according to tocilizumab is administrated by intravenous or sub cutaneous
To compare vitamin B12 serum level (in pmol/L) variation between: infection with tocilizumab / relapse AI/ID with or without tocilizumab / remission state with tocilizumab | from enrollment to the 3 years of the patient's participation
  change of serum level of vitamin B12 (in pmol/L) between sample performed at inclusion and
  * sample performed at Infection without tocilizumab and at remission state with tocilizumab
  * sample performed at relapse AI/ID without tocilizumab and at remission state with tocilizumab
  * sample performed at relapse AI/ID with or without tocilizumab
To study presence of a vitamin B12 serum level (in pmol/L) greater than upper laboratory bound if infection or relapse AI/ID (without tocilizumab) and to compare objectives cited in 2 according to this serum level. | from enrollment to the 3 years of the patient's participation
  Vitamin B12 serum level (in pmol/L) and the presence of serum level of vitamin B12 greater than upper laboratory bound (at University hospital at Clermont fd the normal range are between 178-584 pmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Marc RUIVARD, Pr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No